CLINICAL TRIAL: NCT00094796
Title: Evaluation of Rosiglitazone in Reversing Metabolic Defects of Pre-Diabetes and Type 2 Diabetes Mellitus
Brief Title: Rosiglitazone to Reverse Metabolic Defects in Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050009; 05-H-0009
Record Dates: First submitted 2004-10-22; First posted 2004-10-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-09-03

CONDITIONS: Diabetes Mellitus, Type II; Insulin Resistance
Keywords: Insulin Resistance; Brachial Artery Reactivity; Endothelial Progenitor Cells; Metabolic Stress Test; Mitochondrial Function; Type 2 Diabetes; T2DM; Pre-Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Glucose Intolerance

INTERVENTIONS:
Procedure: Exercise cardiopulmonary metabolic testing
Procedure: Skeletal muscle biopsy
Procedure: Brachial artery reactivity testing

SUMMARY:
This study will examine whether the anti-diabetes medicine rosiglitazone can safely and effectively reverse the early problems of type 2 diabetes and delay the onset of disease in people with pre-diabetes. The underlying problem in people with diabetes or pre-diabetes is insulin resistance (lowered sensitivity to insulin) resulting in poor glucose (sugar) regulation. Rosiglitazone improves the body's sensitivity to insulin.

Patients 21 years of age and older who have type 2 diabetes or who are pre-diabetic (glucose intolerant/insulin resistant) may be eligible for this study. Candidates are screened with a medical history, physical examination, blood tests, echocardiography (heart ultrasound), exercise test, brachial artery reactivity test (see below), and possibly a muscle biopsy.

Participants take one rosiglitazone tablet daily by mouth for 2 weeks. The dose is then increased to two tablets daily for another 2 weeks and then to 4 tablets daily for the remainder of the 12-week treatment period. In addition to treatment, patients undergo the following tests and procedures:

* Resting and exercise metabolic testing: The amount of oxygen taken in and carbon dioxide exhaled during breathing is measured while the patient rests in a chair and then while he or she exercises on a stationary bicycle or treadmill. Both at rest and during exercise, the patient wears a facemask that measures the amount of oxygen used. During exercise, heart rate is monitored with electrodes on the chest, arms, and thighs. The exercise test is repeated three times, once to become familiar with the test, again the next day to measure exercise capacity, and again 3 days later. The third test is less strenuous and is optional.
* Muscle biopsy (optional): A small area of skin over a calf muscle is numbed with a local anesthetic and a 1-inch incision is made over the muscle. A small amount of muscle tissue is taken and the incision is closed with stitches.
* Brachial reactivity study: This ultrasound study tests how well the patient's arteries widen. The subject rests on a bed for 30 minutes. An ultrasound measuring device is placed over the artery just above the elbow. The size of the artery and blood flow through it are measured before and after inflating a pressure cuff around the forearm. The pressure cuff stops the flow of blood to the arm for a few minutes. After a 15-minute rest, a nitroglycerin tablet (medicine that causes blood vessels to relax) is placed under the patient's tongue. Before and 3 minutes after the nitroglycerin is given, the size of the artery and blood flow through it are measured again.
* Blood samples: Blood samples are collected at the beginning and end of the study and at study visits in between.
* Study visits: Patients come to the Clinical Center biweekly or monthly for a follow-up history, physical examination, and blood tests. At the end of the3-month treatment period, they receive recommendations about possible treatment modifications to best maintain glucose tolerance. Their physicians are informed of how their blood sugar was controlled. Six months after completing the study, patients undergo a final study evaluation and blood tests, and are then invited to return for yearly checkups after that.

DETAILED DESCRIPTION:
The majority of insulin resistant individuals (predominantly individuals with type 2 diabetes - T2DM) develop a disproportionate incidence of cardiovascular disease burden including hypertension, coronary artery disease, peripheral vascular disease and heart failure. The underlying pathophysiology is multifactorial but is primarily driven by insulin-resistance mediated regulatory events. These include augmented oxidative stress, upregulation of pro-inflammatory and anti-thrombotic signaling pathways, detrimental effects of advanced glycosylation end-products and perturbations in lipid and fatty acid metabolism. Evidence is emerging to support a role of perturbed mitochondrial respiratory regulation and subsequent endothelial dysfunction as early events in the insulin-resistance syndrome. These in turn, are proposed to result in the subsequent development of the cardiovascular clinical sequelae.

In the last few years, pharmacologic compounds have been developed that directly modulate insulin resistance/sensitivity. Activation of the peroxisome proliferator-activated receptor (PPAR) family of transcription factors has been shown to augment insulin sensitivity. Agents that activate numerous PPAR family members, i.e. pan-PPAR agonists and PPAR gamma (PPAR gamma) specific agonists, promote improved insulin sensitivity. Whether these compounds modify the underlying mitochondrial and endothelial pathophysiology, with the potential of preventing progression of cardiovascular disease in insulin-resistant subjects has not been systematically investigated.

The hypothesis intrinsic to this proposal is that PPAR activation will improve mitochondrial respiratory and endothelial cell function in parallel with improved insulin sensitization in insulin-resistant and T2DM subjects. The primary objective of this study is to establish the effects of the PPAR gamma agonist (rosiglitazone) on exercise-modulated cardiopulmonary-metabolic function (functional measures of mitochrondrial respiratory function) in insulin resistant and T2DM subjects that are either naive to hypoglycemic therapy or are on current therapy with other established classes on anti-diabetic agents with or without associated cardiovascular disease. As secondary end points we will evaluate numerous biological assays of skeletal muscle mitochondrial function, endothelial function and changes in parameters of insulin sensitivity. These include: 1) skeletal muscle mitochondrial respiration, 2) skeletal muscle expression profiles of genes encoding mitochondrial biogenesis program and mitochondrial respiratory control, 3) brachial artery reactivity, 4) endothelial progenitor cell number and colony-forming capacity, 5) monocyte gene expression profiling to evaluate insulin and inflammatory-mediator regulatory events and 6) serological evaluation in change in insulin sensitivity and inflammation. The study is designed as a phase II clinical trial where subjects will receive rosiglitazone for three months duration. Baseline and 3 month laboratory studies will include: 1) rest and exercise cardiopulmonary metabolic testing; 2) skeletal muscle biopsy for mitochondrial function and gene expression profiling analysis, 3) brachial artery reactivity testing and 4) serological and blood cell sampling to determine biochemical, cellular and genomic perturbations in response to insulin-sensitization therapy in this cohort.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults older than 21 years.

Subjects must either have:

1. Insulin resistance as defined by a fasting blood sugar of greater than 110mg/dl and less than 126 mg/dl and confirmed with the QUICKI test.
2. or the diagnosis of T2DM with a HBA1c less than 9%, a fasting insulin level of greater than 6 UIU/ml and a fasting blood glucose level of greater than 125 mg/dl if not on anti-diabetic therapy.

   Subject understands protocol and provides written, informed consent

   Patients must demonstrate the capacity for a near maximal to maximal effort on a treadmill as measured by exercise ventilatory threshold. This will be measured by achieving a peak respiratory exchange ratio greater than or equal to 1.00 during the initial and final peak VO2 exercise tests.

   EXCLUSION CRITERIA:

   Significant structural heart disease (e.g. hypertrophic or dilated cardiomyopathy, valvular heart disease) as determined by echocardiography or unstable coronary disease within the last 3 months.

   Uncontrolled hypertension.

   History of Heart Failure.

   Left ventricular ejection fraction less than 55% as measured by screening echocardiogram.

   Subject physically unable to perform treadmill exercise due to neurologic or orthopedic conditions.

   Insulin-dependent diabetes mellitus or current use of thiazolidinediones

   History of adverse events on thiazolidinedione therapy

   Women of childbearing age unless recent pregnancy test is negative.

   Lactating women.

   Serum creatinine greater than 2.5 mg/dl

   Liver transaminase levels greater than 2.5 x upper limit of normal

   History of cancer in the last 5 years

   History of treatment for any illness with stem cell transplantation

   Active inflammatory disease

   Enrollment in a any drug studies within the last 30 days

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2004-10-20; Study Completion 2008-09-03

PRIMARY OUTCOMES:
Peak VO(2) after 3 months of rosiglitazone therapy compared with baseline VO(2) max.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Medical College of Virginia, Richmond, Virginia

REFERENCES:
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527